CLINICAL TRIAL: NCT07230353
Title: A Phase 1b, Open-label, Dose-Escalation Trial to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Plamotamab in Participants With Rheumatoid Arthritis
Brief Title: A Phase 1b Open-label Study to Evaluate Safety in Participants With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XmAb13676-06
Record Dates: First submitted 2025-10-01; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, Arthritis Rheumatoid, Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dose Escalation (Experimental): XmAb 13676 administered SC
  Interventions: Biological: XmAb13676

INTERVENTIONS:
Biological: XmAb13676 — Biological

SUMMARY:
The purpose of this study is to determine the safety and tolerability of XmAb13676 in patients with rheumatoid arthritis. Participants will be given XmAb13676 subcutaneously (SC) by injection under the skin.

DETAILED DESCRIPTION:
This is a Phase 1b study to determine the safety, tolerability, pharmacokinetic (PK), and pharmacodynamics (PD), and immunogenicity of XmAb13676 in adult participants with moderately to severely active RA. This is an open label dose optimization trial with approximately 47 participants assigned to different dose escalation cohorts.

ELIGIBILITY:
Inclusion Criteria: Adult participants with moderately to severely active RA.

* Documented diagnosis of RA and meeting the 2010 American College of Rheumatology/European Alliance of Associations for Rheumatology classification criteria for RA at least 3 months prior to screening
* Inadequate response to, loss of response to, or intolerance to available RA therapies.
* Stable doses of RA medications prior to screening
* Use of highly effective methods of contraception

Exclusion Criteria:

* Major surgery within 12 weeks prior to screening or planned within 12 months after dosing
* Recurrent infections or active clinically significant infection
* Active or untreated latent tuberculosis
* Cancer or history of cancer or lymphoproliferative disease within the previous 5 years
* Uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease

Note: Additional, more specific inclusion/exclusion criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Primary | Through Week 52
  Percentage of participants with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Secondary | Through Week 52
  Serum concentration of plamotamab

CONTACTS AND LOCATIONS:
Overall Officials: Mark Osterman, MD, MS, Study Director — Xencor, Inc.
Locations (4):
- Georgia (2):
  - Arensia Research Clinic, Tbilisi
  - Xencor Investigative Site, Tbilisi
- Arensia Research Clinic, Chisinau, Moldova
- Xencor Investigative Site, Auckland, New Zealand